CLINICAL TRIAL: NCT00822536
Title: Optimal Duration of Dual Antiplatelet Therapy After Drug Eluting Stent (DES) Implantation
Brief Title: Optimal Duration of Dual Antiplatelet Therapy After Drug-eluting Stent Implantation
Acronym: OPTIDUAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071210
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease; Stent Thrombosis; Myocardial Ischemia
Keywords: Drug-eluting stent; Clopidogrel; Stent thrombosis; Myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bi therapy : aspirin/ clopidogrel
  Interventions: Drug: Aspirin and Clopidogrel
- 2 (Active Comparator): Monotherapy: aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin and Clopidogrel — Aspirin <= 325 mg/j Clopidogrel = 75 mg /j
  Other Names: Aspirin: acid acetylsalycilic; Clopidogrel: plavix
  Arms: 1
Drug: Aspirin — Aspirin : <= 325 mg/j
  Other Names: Aspirin: acid acetylsalycilic
  Arms: 2

SUMMARY:
To compare treatment with aspirin alone versus the combined antiplatelet treatment aspirin and clopidogrel after 12 months of combined antiplatelet treatment following drug-eluting stent (DES) implantation.

DETAILED DESCRIPTION:
Drug-eluting stents (DES) substantially reduce restenosis compared with bare metal stents and represent a significant advance in percutaneous coronary interventions (PCIs). Accordingly, DES have been rapidly adopted into practice and are currently used in the majority of PCI procedures. Despite their rapid acceptance, DES are not without limitations. In particular, patients who receive DES (like those who receive conventional bare metal stents) remain at risk of a 1% to 2% incidence of stent thrombosis, which is often associated with devastating consequences like death or myocardial infarction. Understanding and eliminating mediators of stent thrombosis are thus important goals for optimizing the clinical benefits of DES. Delayed endothelial coverage after DES implantation has been demonstrated and is thought to prolong the window of vulnerability to stent thrombosis. Consequently, current recommendations for DES are: dual antiplatelet therapy for at least 12 months in patients at low risk of bleeding, especially with " off-label " use. Because of rare but severe very late stent thrombosis, the dual antiplatelet therapy is more and more prescribed in clinical practice for several years.But it has been clearly demonstrated that the combination of aspirin and clopidogrel (the thienopyridine the most used) significantly increase the rate of severe and moderate bleedings when compared to aspirin alone. This is important if we consider the possibility or the necessity to prolong the combined antiplatelet therapy after stent implantation.ProposalTo compare treatment with aspirin alone versus the combined antiplatelet treatment with aspirin and clopidogrel after 12 months of combined antiplatelet treatment after DES implantation

NB : On the decision of the sponsor, the latest patient monitoring was advanced to September 30, 2014 instead of January 2015.

ELIGIBILITY:
Inclusion can be done either after stenting or 12 months later :

A: Patients admitted for DES implantation can be selected. After 12 months of bi therapy, they will be randomized

B: patients who have got a DES implantation 12 months before can be selected and randomised

Inclusion criteria:

* Patients on aspirin and clopidogrel therapy at 12 months after DES implantation
* Informed, written consent by the patient

Exclusion criteria:

* DES in left main coronary artery
* Oral anticoagulation therapy with coumadin derivatives
* Active bleeding; bleeding diathesis; history intracranial bleeding
* Known allergy or intolerance to the study medications: aspirin and clopidogrel
* Pregnancy (present, suspected or planned) or positive pregnancy test (In women with childbearing potential a negative pregnancy test is mandatory)
* Patient's inability to fully comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1798 (Actual)
Dates: Start 2009-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite criteria : death, non fatal myocardial infarction, non fatal stroke and severe bleeding | At each visit (every 6 months) with Follow-up of 3 years

SECONDARY OUTCOMES:
Death | At each visit (every 6 months) with Follow-up of 3 years
Non fatal myocardial infarction | At each visit (every 6 months) with Follow-up of 3 years
Non fatal stroke | At each visit (every 6 months) with Follow-up of 3 years
Severe bleeding | At each visit (every 6 months) with Follow-up of 3 years
Stent thrombosis (ARC définition) | At each visit (every 6 months) with Follow-up of 3 years
Target lesion revascularization | At each visit (every 6 months) with Follow-up of 3 years
Moderate bleeding (ISTH definition) | At each visit (every 6 months) with Follow-up of 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gérard HELFT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital la Pitié Salpêtrière Institut de Cardiologie, Paris, France

REFERENCES:
- [Derived] Helft G, Steg PG, Le Feuvre C, Georges JL, Carrie D, Dreyfus X, Furber A, Leclercq F, Eltchaninoff H, Falquier JF, Henry P, Cattan S, Sebagh L, Michel PL, Tuambilangana A, Hammoudi N, Boccara F, Cayla G, Douard H, Diallo A, Berman E, Komajda M, Metzger JP, Vicaut E; OPTImal DUAL Antiplatelet Therapy Trial Investigators. Stopping or continuing clopidogrel 12 months after drug-eluting stent placement: the OPTIDUAL randomized trial. Eur Heart J. 2016 Jan 21;37(4):365-74. doi: 10.1093/eurheartj/ehv481. Epub 2015 Sep 12. PMID 26364288
- [Derived] Helft G, Le Feuvre C, Georges JL, Carrie D, Leclercq F, Eltchaninoff H, Furber A, Prunier F, Sebagh L, Cattan S, Cayla G, Vicaut E, Metzger JP. Efficacy and safety of 12 versus 48 months of dual antiplatelet therapy after implantation of a drug-eluting stent: the OPTImal DUAL antiplatelet therapy (OPTIDUAL) trial: study protocol for a randomized controlled trial. Trials. 2013 Feb 21;14:56. doi: 10.1186/1745-6215-14-56. PMID 23433461